CLINICAL TRIAL: NCT03624894
Title: Suitability of Intraoral Impressions for Assessment of Wear of Teeth and Restorative Materials Over 60 Months Using the Replica Method and 3-D Laser Equipment.
Brief Title: Intraoral Impressions for Assessment of Wear of Teeth and Restorative Materials.
Acronym: GIC
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: I.R.C.C.S Ospedale Galeazzi-Sant'Ambrogio (Other)
Responsible Party: Sponsor
Other Study IDs: GIC
Record Dates: First submitted 2018-03-13; First posted 2018-08-10 (Actual); Last update posted 2018-08-10 (Actual); Status verified 2018-08

CONDITIONS: Wear, Tooth; Wear, Occlusal; Wear, Restoration
Keywords: oral impressions; glassionomer cements; dental restorations; dental wear
MeSH Terms: conditions — Tooth Wear; Tooth Attrition | interventions — Inosine Monophosphate

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients that undergo a dental restorations: Patients that undergo a dental restorations independently from the present study
  Interventions: Other: impression

INTERVENTIONS:
Other: impression — common polyvinylsiloxane oral impression

SUMMARY:
Suitability of intraoral impressions for assessment of wear of teeth and restorative materials over 60 months, using the gypsum replica method and 3-D laser scanning: perspective clinical and laboratory evaluation.

DETAILED DESCRIPTION:
The study will assess suitability of intraoral impressions for assessment of wear of artificial dental restorative materials over 60 months. Subjects are recruit from patients that undergo a dental restorations independently from the present study. The sample size of n=65 would enable detection of differences in material and tooth wear greater than 10-13% from the baseline volume of teeth, when compared with volumes of teeth obtained from impressions taken at follow-ups, with the power of 0.8 and for the significance level of p=0.05. Paired t-test or a Wilcoxon signed-rank test is implemented depending on the distribution of the variables, for primary aim of evaluating suitability of polyvinylsiloxane dental impression for determination of wearing of teeth and restorative materials.

Paired t-test for each sub-score or a Wilcoxon-signed rank test is implemented, depending on the distribution of the variables, for secondary aims. Then, if variables are considered also as categorical, a Mc Nemar test for each sub-score will be suggested

ELIGIBILITY:
Inclusion Criteria:

1. Subject ≥18 years.
2. Subjects with restorative treatments on vital teeth in posterior molar region. Will be considered at most one reconstruction per side.
3. Restorations limited to two surfaces (Black's Class II) with one proximal cavity, in occlusion. Max 1 restoration will be included each oral side (right or left).
4. Favorable and stable occlusal relationship between the remaining teeth.
5. Subject must be reliable, cooperative, and in the opinion of the Investigator, likely to be compliant with study procedures.
6. Subject provides written informed consent signed and dated prior to entering the study.

Exclusion Criteria:

Inclusion and exclusion criteria

Inclusion criteria

1. Subject ≥18 years.
2. Subjects with restorative treatments on vital teeth in posterior molar region. Will be considered at most one reconstruction per side.
3. Restorations limited to two surfaces (Black's Class II) with one proximal cavity, in occlusion. Max 1 restoration will be included each oral side (right or left).
4. Favorable and stable occlusal relationship between the remaining teeth.
5. Subject must be reliable, cooperative, and in the opinion of the Investigator, likely to be compliant with study procedures.
6. Subject provides written informed consent signed and dated prior to entering the study.

Exclusion criteria

1. Subject with full dentures or crowns and bridges in occlusal contact with teeth indicated for restorative treatment.
2. Absence of occlusal contact.
3. Subject has a history of drug abuse, addiction to medication or alcohol abuse within the previous year.
4. Pulp exposure during restorative procedure or unvital teeth.
5. Known unavailability of subject for recall Visit(s).
6. Allergy to any ingredient of impression material.
7. Severe bruxism.
8. Subject with clinically significant or unstable medical or physiological condition.
9. Female subject is pregnant or lactating or intends to become pregnant during the course of the study.
10. Subject is not willing to participate in the study or not able to understand the content of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects are recruit from patients that undergo a dental restorations independently from the present study
Sampling Method: Non-Probability Sample
Enrollment: 33 (Actual)
Dates: Start 2016-02-01 (Actual); Primary Completion 2021-02-01 (Estimated); Study Completion 2021-11-16 (Estimated)

PRIMARY OUTCOMES:
Wear of teeth and materials of restorations | 5 years
  3D models will be obtained from intraoral impressions taken at baseline, at 3 and at 5 years fo follow-up. 3D models obtained at different times will be compared by a 3D software (Aadva LabScan Software, GC Corporation, Japan), able to overlap the volumes and identify all areas where surfaces have been worn. The software is able to create graphical images of the occurred wear, but also to numerically quantify the volume lost due to wear. The software is able to evaluate differences till 0,001 mm, but for this study the limit for precision had been set to 0,01 mm.

SECONDARY OUTCOMES:
Level of wear of different restorative materials | 5 years
  The 3D evaluation of wear will identify the entity of wear for different substrates, and different behaviour of dental material will be possibly highlighted. Is it more than possible that under the same biting forces, different materials will show different wear, revealing which of them will be more suitable for long term, successful, dental restoration.

IPD SHARING:
Plan to Share IPD: Undecided